CLINICAL TRIAL: NCT05488041
Title: Characteristics of Anal Manometry Examination in Patients With Ulcerative Colitis (UC) in Remission With Anorectal Symptoms in a New Disease Compared to a Disease of Many Years
Brief Title: Anal Manometry Examination in Patients With Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Meir Medical Center (Other); Nazareth Hospital (Other)
Responsible Party: Principal Investigator, Vered Richter, Principal Investigator, Assaf-Harofeh Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0232-21-ASF
Record Dates: First submitted 2021-11-16; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC patients with anorectal symptoms (Experimental): Patients with ulcerative colitis in remission who have anorectal symptoms will undergo an anal manometry test to characterize these symptoms.
  Interventions: Procedure: Performing anorectal manometry
- UC patients without anorectal symptoms (Active Comparator): Patients with ulcerative colitis in remission without anorectal symptoms will undergo an anal manometry test to characterize their anorectal function and to compare to those with symptoms
  Interventions: Procedure: Performing anorectal manometry

INTERVENTIONS:
Procedure: Performing anorectal manometry — Anorectal manometry is a safe, low-risk procedure and is unlikely to cause any pain, colorectal perforation is very rare. Seven cases have been published in four reports.
  * Anorectal Manometry - NY Gastroenterology Associates n.d. https://www.gastroenterologistnewyork.com/preparing-for-procedure/anorectal-manometry/ (accessed July 14, 2021).
  * Bionda M, Lenglinger J, … AH-J of E, 2020 undefined. Closure of Large Rectal Iatrogenic Perforation by Endoscopic Suture Device: Go for it. BorisUnibeCh 2020;01:13-5. https://doi.org/10.48350/151165.

SUMMARY:
Inflammatory bowel diseases (IBD), which include Crohn's disease (CD) and ulcerative colitis (UC), are chronic immune-related diseases. IBD symptoms frequently overlap with symptoms of functional GI disorders such as irritable bowel syndrome (IBS) and defecatory disorders, and these symptoms are common in patients with active disease, and also in quiescent disease. Underdiagnosis of abnormal anorectal function may result in an inappropriate escalation of IBD therapy. In this study, the investigators aim to evaluate if damage from chronic inflammation in UC results in anorectal damage such as hypersensitive, hyperactive, poorly compliant rectum, and hypotensive sphincter. If this is the case, early aggressive treatment of the disease is needed.

Another important point in this study is to find out which of the anorectal symptoms are due to a hypersensitive, hyperactive, and poorly compliant rectum and not due to mucosal inflammation. The diagnosis of abnormal anorectal function via manometry may help to give the appropriate treatment, such as biofeedback or pharmacological treatment such as loperamide or tricyclic anti-depressants. This may avoid escalation or replacing effective IBD therapy unnecessarily.

DETAILED DESCRIPTION:
The study will include patients with ulcerative colitis in clinical, laboratory, and endoscopic remission, and with one of the following symptoms: Urgency, fecal incontinence, incontinence to gas, tenesmus, rectal discomfort, rectal pain, excessive straining and incomplete evacuation.

Patients that will not be included: patients after ileal pouch-anal anastomosis (IPAA), and patients with colonic stenosis that could not be passed with an endoscope.

Patients will undergo an anorectal manometry test and the results will be compared to a control group that will include patients with ulcerative colitis in remission without anorectal complaints, as well as to the normal values in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with UC in our clinics who have one of the following symptoms: Urgency, fecal incontinence, incontinence to gas, tenesmus, rectal discomfort, rectal pain, excessive straining, and incomplete evacuation
* A patient who has had a recent colonoscopy/sigmoidoscopy with endoscopic remission defined as Mayo endoscopic score ≤1

Exclusion Criteria:

* Patient after ileal pouch-anal anastomosis surgery (IPAA)
* Patients with colonic stenosis that did not allow endoscopic passage and did not undergo an endoscopic evaluation prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Defecation disorders in patients with UC | Two years
  To evaluate the rate and types of defecation disorders in patients with UC in remission as examined by anorectal manometry (ARM), and to examine the correlation between these anorectal pathologies and disease duration in years.

SECONDARY OUTCOMES:
To examine a possible correlation between the findings in anal manometry and other disease parameters, clinical, laboratory, and histological characteristics. | Two years
  The investigators will examine a possible correlation between defecation disorders in patients with UC in remission to the following parameters: disease characteristics: disease extension, presence of stenosis, presence of anal fissure or hemorrhoids, levels of CRP and calprotectin, presence of extra-intestinal manifestations; to symptoms such as the number of defecations per day, the texture of stool according to Bristol, exertion effort, feeling of emptiness, tenesmus, use of laxatives / anti-diarrhea medication, use of leakage pads; to findings in biopsies taken from the last colonoscopy/sigmoidoscopy.
  A comparison will be made to a control group of UC patients in remission without anorectal symptoms, as well as to the normal values in the literature

CONTACTS AND LOCATIONS:
Overall Officials: Vered Richter, Dr, Principal Investigator — Shamir (Assaf-Harofeh MC)
Locations (1):
- Shamir Medical Center (Assaf Harofeh), Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No
All patient data will be securely stored at the medical center